CLINICAL TRIAL: NCT02403622
Title: Safety of Fecal Microbiota Transplantation: OpenBiome Outcomes and Longitudinal Follow-up (STOOL) for Recurrent Clostridium Difficile Infection
Brief Title: Safety of FMT: OpenBiome Outcomes and Longitudinal Follow-up (STOOL) for Recurrent Clostridium Difficile Infection
Acronym: STOOL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: for futility
Sponsor: Microbiome Health Research Institute (Other)
Collaborators: Brown University (Other); Edward Hospital (Other); Indiana University (Other); Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1410006671
Record Dates: First submitted 2015-03-06; First posted 2015-03-31 (Estimated); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Clostridium Difficile

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention: Fecal Microbiota Preparation (Experimental): Open label single arm Dosage form: Screened human donor stool, sourced from human-derived microbes generated by healthy, screened donors.
  Route of administration: either colonoscopic/sigmoidoscopic FMT or retention enema FMT Dosing Regimen: 250 mL x 1 dose. In the event of a clinical non-response, a repeat single 250 mL dose will occur from a different donor
  Interventions: Drug: Fecal Microbiota Preparation

INTERVENTIONS:
Drug: Fecal Microbiota Preparation — Frozen processed human fecal material for treating recurrent Clostridium difficile infections.

SUMMARY:
The overarching objective of this study is to address the knowledge gap regarding the short-term and long-term safety of fecal microbiota transplants (FMT). The design will be a prospective, open-label, multi-center longitudinal cohort study to assess the short- and long-term safety of FMT as well as the clinical resolution of diarrhea among 150 patients with 3 or more episodes of clostridium difficile infection (CDI defined as 3 unformed stools over 24 hours for 2 consecutive days and either a positive stool test for CDI or pseudomembranes on colonoscopy/sigmoidoscopy). Subjects will be adult outpatients referred to one of the study centers after at least three recurrent episodes of CDI and previous treatment with at least one 10-day course of oral vancomycin or fidaxomicin. After FMT by colonoscopy/sigmoidoscopy or enema, patients will be followed prospectively and monitored for clinical resolution and adverse events at: 3 days (telephone), 3 weeks (clinical assessment), 8 weeks (telephone), 6 months (telephone), and 12 months (telephone) after FMT. Subjects who recur will be offered a second FMT by colonoscopy with a different donor. Microbiome analysis will be conducted from stool samples at baseline and each of the 5 follow-up intervals.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18-75 years old)
* Outpatient
* Third or further documented CDI episode and
* Unable to maintain CDI cure after standard therapy with oral vancomycin or fidaxomicin

  * Previous treatment with at least one course of tapered/pulse vancomycin or
  * Inability to taper or stop vancomycin or fidaxomicin without developing diarrhea requiring antibiotic therapy.
* Improvement of CDI symptoms on vancomycin or fidaxomicin

Exclusion Criteria:

* Unable to comply with study follow-up procedures at discretion of MD
* Unable to provide informed consent at discretion of MD
* Participating in another clinical trial
* Pregnant or nursing currently or planned pregnancy in next 1 year
* Evidence of toxic megacolon or gastrointestinal perforation
* Peripheral white blood cell count >30 x 10^9/L and/or temperature >38 degrees Celsius
* Admission to an intensive care unit within prior 7 days for any reason
* Previously undergone FMT
* Severely immunocompromised patients

  * HIV infection (any CD4 count)
  * AIDS-defining diagnoses
  * Inherited/primary immune disorder
  * Immunosuppressant medications:
* Current or recent (<3 months) treatment with anti-neoplastic agents
* Current or recent (<3 months) treatment with calcineurin inhibitors (tacrolimus, cyclosporine)
* Current or recent (<3 months) treatment with mycophenolate mofetil
* Current or recent (<3 months) treatment with monoclonal antibodies to B and T-Cells, anti-TNF, glucocorticoids, antimetabolites (azathioprine, 6-mercaptopurine)
* Neutropenia with absolute neutrophil count (ANC) <0.5 x 10^9/L
* Active gastroenteritis due to infectious cause other than CDI
* Short gut syndrome
* Colostomy
* Ascites
* End-stage liver disease
* Untreated, in-situ colorectal cancer
* Irritable bowel syndrome
* Inflammatory bowel disease including Crohn's disease and ulcerative colitis
* Microscopic colitis including collagenous colitis and lymphocytic colitis
* Severe food allergy (anaphylaxis) that cannot be confirmed as having been excluded from a donor's diet within the five days prior to donation
* Anorectal disorder/severe rectal sphincter tone abnormality or inability to retain enema material
* Unable or unwilling to tolerate colonoscopy/sigmoidoscopy, colonoscopy prep, or enema for any reason at discretion of MD
* Severe underlying disease that the patient is not expected to survive for the subsequent 12 months at the discretion of the MD.
* Any conditions for which, in opinion of MD, the treatment may pose a health risk

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Edward Hospital, Naperville, Illinois
  - IU University Hospital, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 17 participants enrolled (signed consents) across four sites during the period between March 27, 2015 and October 4, 2017.
Pre-assignment Details: Two enrolled participants withdrew from the study prior to intervention.
Groups:
- Intervention: Fecal Microbiota Preparation: Open label single arm Dosage form: Screened human donor stool, sourced from human-derived microbes generated by healthy, screened donors.
  Route of administration: either colonoscopic/sigmoidoscopic FMT or retention enema FMT Dosing Regimen: 250 mL x 1 dose. In the event of a clinical non-response, a repeat single 250 mL dose will occur from a different donor
  Fecal Microbiota Preparation: Frozen processed human fecal material for treating recurrent Clostridium difficile infections.
Period: Overall Study
Arm/Group | Intervention: Fecal Microbiota Preparation
Started | 15
Completed | 13
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Baseline population includes all participants who had enrolled (signed consent) in the study.
Arm/Group | Intervention: Fecal Microbiota Preparation
Number analyzed (Participants) | 17
Age, Customized [Count of Participants; unit: Participants]
  Age: 18 to 35 years | 0
  Age: 35 to 55 years | 8
  Age: 55 to 75 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Short-term Safety of FMT as Measured by Absence or Presence of Related Serious Adverse Events
Description: Determine the short-term safety of FMT for the prevention of further CDI recurrence. Short-term safety was measured by absence or presence of related serious adverse events
Time Frame: < 6 weeks post FMT
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: Fecal Microbiota Preparation
Number analyzed (Participants) | 15
Participants | 0

2. Primary Outcome: Long-term Safety of FMT as Measured by Absence or Presence of Adverse Events
Description: Determine the long-term safety of FMT for the prevention of further CDI recurrence
Time Frame: > 6 weeks to 1 year post FMT
Population: Data were not collected therefore could not be reported.
Arm/Group | Intervention: Fecal Microbiota Preparation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: As outlined in the protocol, safety data were collected up to 12 months post-FMT. Due to study termination, not all participants were followed for the full 12 months, but instead an average of 11.7 months.
Arm/Group | Intervention: Fecal Microbiota Preparation
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention: Fecal Microbiota Preparation (N=15)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1)
Gastrectomy (Surgical and medical procedures) | 1 (1)
Pancreatectomy (Surgical and medical procedures) | 1 (1)
Splenectomy (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention: Fecal Microbiota Preparation (N=15)
Abdominal Pain (Gastrointestinal disorders) | 7 (8)
Bloating/Distention (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (7)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Flatulence (Gastrointestinal disorders) | 6 (8)
Nausea (Gastrointestinal disorders) | 1 (1)
Increase in bowel movements (Gastrointestinal disorders) | 1 (1)
Incontinence (Gastrointestinal disorders) | 1 (1)
Knee Replacement (Surgical and medical procedures) | 1 (1)
Laparoscopy (Surgical and medical procedures) | 1 (1)
UTI (Infections and infestations) | 5 (6)
CDI (Infections and infestations) | 1 (1)
Stroke (Vascular disorders) | 1 (1)
Weight gain (Metabolism and nutrition disorders) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 1 (1)
Thyrotoxicosis (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Graves' Disease (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Fatigue and malaise (General disorders) | 1 (1)
Allergies (Immune system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
5th Metatarsal fracture (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-03): https://cdn.clinicaltrials.gov/large-docs/22/NCT02403622/Prot_SAP_000.pdf